CLINICAL TRIAL: NCT02033551
Title: An Extension Study to Evaluate the Safety of Veliparib as Single Agent Therapy or in Combination With Chemotherapy in Subjects With Solid Tumors
Brief Title: A Study Evaluating Veliparib as a Single Agent or in Combination With Chemotherapy in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-144; 2013-003137-16 (EudraCT Number)
Record Dates: First submitted 2014-01-08; First posted 2014-01-13 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer; Ovarian Cancer; Colon Cancer; Lung Cancer; Gastric Cancer; Solid Tumors
Keywords: Gastric Cancer; Lung Cancer; PARP Inhibitor; Ovarian Cancer; Solid Tumors; Breast Cancer; Colon Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Colonic Neoplasms; Lung Neoplasms; Stomach Neoplasms | interventions — veliparib; Carboplatin; Paclitaxel; IFL protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A - Veliparib Monotherapy (Experimental): Subjects in this arm will be dosed with Veliparib continuous dosing.
  Interventions: Drug: Veliparib
- Arm B - Veliparib in Combination with Carboplatin & Paclitaxel (Experimental): Subjects enrolled will receive Veliparib in combination with Carboplatin and Paclitaxel and have an option to move to Veliparib monotherapy.
  Interventions: Drug: Veliparib; Drug: Carboplatin; Drug: Paclitaxel
- Arm C Veliparib in Combination with Modified FOLFIRI (Experimental): Subjects will be given Veliparib in combination with modified FOLFIRI. The subject will have the opportunity to receive Veliparib as monotherapy.
  Interventions: Drug: Veliparib; Drug: FOLFIRI

INTERVENTIONS:
Drug: Veliparib
  Other Names: ABT-888
Drug: Carboplatin
  Arms: Arm B - Veliparib in Combination with Carboplatin & Paclitaxel
Drug: Paclitaxel
  Other Names: Taxol
  Arms: Arm B - Veliparib in Combination with Carboplatin & Paclitaxel
Drug: FOLFIRI — combination of Fluorouracil, leucovorin and irinotecan
  Arms: Arm C Veliparib in Combination with Modified FOLFIRI

SUMMARY:
This is an extension study to evaluate the safety of Veliparib monotherapy or in combination with Carboplatin plus Paclitaxel or modified Folinic Acid/Fluorouracil/Irinotecan (FOLFIRI) in subjects with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Must have confirmed solid malignancy that is metastatic, and standard curative measures or other therapy that may provide clinical benefit do not exist or are no longer effective.
* For Veliparib monotherapy (must have tumor with defects in DNA repair mechanisms (BRCA mutation or high grade ovarian cancer or solid tumors for combination therapy.
* If the subject has known brain metastases must have clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function and no evidence of Central Nervous System (CNS) disease progression as determined by comparing a computed tomography (CT) scan or magnetic resonance imaging (MRI) scan performed during screening to a prior scan performed at least 4 weeks earlier and provided that the subject is asymptomatic, has no evidence of cavitation or hemorrhage, and does not require corticosteroids (must have discontinued steroids at least 3 months prior to study drug administration).
* Subject must have adequate bone marrow, renal and hepatic function per local laboratory reference range.

Exclusion Criteria:

* Subject has a clinically significant and uncontrolled major medical condition(s) including but not limited to:
* Uncontrolled seizure disorder, including focal or generalized seizure within the last 12 months;
* Uncontrolled nausea/vomiting/diarrhea;
* Active uncontrolled infection;
* Symptomatic congestive heart failure;
* Unstable angina pectoris or cardiac arrhythmia;
* Psychiatric illness/social situation that would limit compliance with study requirements;
* Any medical condition, which in the opinion of the study investigator, places the subject at an unacceptably high risk for toxicities.
* Subjects who have hypersensitivity to Carboplatin, Paclitaxel or Cremophor should be excluded from arm B.
* Subject has received any of the following anti-cancer therapies 21 days prior to the first dose of study drug or a biologic agent for anti-neoplastic intent within 30 days prior to the first dose of study drug.
* Subject who requires parenteral nutrition, tube feeding or has evidence of a partial bowel obstruction or perforation within 28 days prior to study drug.
* The subject has had another active malignancy within the past 3 years except for any cancer in situ that the Principal Investigator considers to be cured.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events | Measured up to 30 days after the last dose of study drug.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Radiographic evaluation at Screening and every 6-9 weeks until the final visit, up to 18 months.
Overall Survival (OS) | Every 3 months after the subject is registered off study up to 2 years post discontinuation or until date of death from any cause, whichever comes first.
Time to Disease Progression (TTP) | Assessed at each visit up to 18 months after the last subject has enrolled in the study.
Progression Free Survival (PFS) | Radiographic evaluation starting from the first day of study drug until documented progression or date of death, whichever comes first, until the subject is registered off study.
Clinical Laboratory Tests | Up to 18 months.
  Hematology, Chemistry, Urinalysis
Electrocardiogram | Up to 18 months.
Tumor Assessment | Up to 18 months.
  A computerized tomography scan to document the size of the tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Shepherd, PhD, Study Director — AbbVie
Locations (5):
- United States (2):
  - Site Reference ID/Investigator# 117416, Scottsdale, Arizona
  - Site Reference ID/Investigator# 117415, San Antonio, Texas
- Netherlands (2):
  - Site Reference ID/Investigator# 117337, Groningen
  - Site Reference ID/Investigator# 117338, Maastricht
- Site Reference ID/Investigator# 117451, Madrid, Spain